CLINICAL TRIAL: NCT02195739
Title: A Retrospective, Real-life Evaluation of the Cardiovascular Disease Risk Associated With Exposure to Pharmacological Smoking Cessation Interventions in a Representative UK Primary Care Patient Population.
Brief Title: Nicotine Replacement Therapy and Cardiovascular Disease
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Research in Real-Life Ltd (Network)
Responsible Party: Sponsor
Other Study IDs: E02311
Record Dates: First submitted 2014-05-14; First posted 2014-07-21 (Estimated); Last update posted 2014-10-01 (Estimated); Status verified 2014-09

CONDITIONS: Smoking Cessation
Keywords: smoking; smoking cessation; cardiovascular disease; pharmacological intervention; UK primary care population; nicotine replacement therapy
MeSH Terms: conditions — Smoking Cessation; Smoking; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Nicotine replacement therapy cohort: Cohort defined as patients in whom nicotine replacement therapy (in any preparation) was initiated at the index smoking cessation attempt as the first recorded smoking cessation intervention.
- Other smoking cessation therapy: Cohort defined as patients in whom other (non-nicotine replacement therapy) smoking cessation pharmacotherapy's were initiated at the index smoking cessation attempt (e.g. bupropion, varenicline) as the first recorded smoking cessation intervention
- Smoking cessation advice cohort: Cohort (control patients) defined as patients whose first recorded smoking cessation intervention involved smoking cessation advice leading to a quit attempt unassisted by pharmacological smoking cessation aids, at the index smoking cessation attempt.

SUMMARY:
The aim of this study is to compare the cardiovascular disease event rate in smokers undertaking pharmacologically unaided smoking cessation attempts (the non-exposed group) with the event rate in smokers attempting smoking cessation assisted by pharmacological interventions - by nicotine replacement therapy (as any, or a combination, of: nasal spray, transdermal patches, inhaler or gum and tablets) or other pharmacological smoking cessation aids (e.g. bupropion [Zyban®] and varenicline [Champix®]) - in a representative UK primary care population.

DETAILED DESCRIPTION:
Preliminary study data have indicated a possible increased cardiovascular disease risk in patients exposed to nicotine replacement therapy compared with controls (i.e. non-nicotine replacement therapy exposed patients) of a magnitude that could not reasonably be accounted for by differences in the cardiovascular risk profile of the two patient groups. Further in-depth studies in this area are warranted.

This retrospective study will compare the cardiovascular disease event risk in a group of smokers undertaking pharmacologically unaided smoking cessation attempts with the event rate in a group of smokers attempting smoking cessation assisted by pharmacological interventions (any of nicotine replacement therapy, bupropion or varenicline) in a representative UK primary care population.

There are three main types of pharmacological interventions currently available for smoking cessation, each of which has demonstrated efficacy when used in conjunction with behavioural support: nicotine replacement therapy, bupropion, and varenicline. Other medications, especially nortryptiline and clonidine, are considered to be effective adjunct therapy in smoking cessation, but they remain second-line options at this time.

Nicotine replacement therapy has been available since the 1980s and bupropion since 2000. Either approach to cessation doubles the chance of achieving abstinence when compared with unsupported quit attempts. After being granted its European licence in 2006, varenicline joined the pharmacological smoking cessation armamentarium. It is the first drug developed specifically for the treatment of tobacco dependence that contains no nicotine, and it triples smokers' chances of quitting compared with unsupported quit attempts.

As the fore-runner, nicotine replacement therapy is the longest-standing of the existing pharmacological smoking cessation interventions currently available. It aims to alleviate nicotine withdrawal symptoms by substituting the nicotine attained through tobacco smoking via alternative means (e.g. nasal sprays, inhalers, gum and tablets, transdermal patches). The various nicotine replacement therapy products available have differing durations of action and allow patients to tailor their nicotine intake according to their particular needs.For example, patches can be used to substitute for background nicotine and gums or tablets can be used to help satisfy urges.

ELIGIBILITY:
Inclusion Criteria:

* The analysis will include an exposure group comprising smokers with no recorded smoking cessation attempts using pharmacological aids in the prior year, whose first recorded smoking cessation intervention was a cessation attempt assisted by either nicotine replacement therapy (using any of, or a combination of products) or another pharmacological smoking cessation intervention (e.g. bupropion, varenicline) at the index date.

Patients must also meet the following inclusion criteria:

* Aged: 18-75 years.
* Have at least one year of up-to-standard baseline data as defined by Clinical Practice Research Datalink (prior to the index smoking cessation attempt) and at least one year of up-to-standard outcome data (following the index smoking cessation attempt) or up-to-standard data up to the time of death if death occurred within the outcome period.

Exclusion Criteria:

Patients will be excluded from the analysis if they:

* Have had exposure to any nicotine replacement therapy or other pharmacological smoking cessation interventions in the baseline period (year prior to the index smoking cessation attempt), and/or
* Switched between types of smoking cessation interventions (i.e. nicotine replacement therapy to other pharmacological smoking cessation interventions or vice versa) during the outcome period(s). Switching between different nicotine replacement therapy products, or use of multiple nicotine replacement therapy products, will be permissible and analysis may involve a comparison of outcomes relative to nicotine exposure over the various outcome periods.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: EXPOSED PATIENTS: include smokers with no recorded smoking cessation attempts using pharmacological aids in the prior year, whose index smoking cessation attempt was assisted by one of the following pharmacological interventions:
  (i) nicotine replacement therapy as any, or a combination, of transdermal patches, nasal spray, gum and tablets, inhaler.
  (ii) Other (e.g. bupropion, varenicline).
  NON-EXPOSED PATIENTS: include smokers with no recorded smoking cessation attempts using pharmacological aids in the prior year, whose index smoking cessation attempt involved receipt of smoking cessation advice that resulted in a quit attempt unaided by pharmacological therapies.
Sampling Method: Non-Probability Sample
Enrollment: 61050 (Actual)
Dates: Start 2013-09; Primary Completion 2014-03 (Actual); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Time to first coronary heart disease diagnosis | 4 weeks
  Analysed using Cox's proportional hazards model. Time from index smoking cessation attempt. Excluding patients with prior coronary heart disease.
Time to first cerebrovascular disease diagnosis. | 4 weeks
  Analysed using Cox's proportional hazards model. Time from index smoking cessation attempt. Excluding patients with prior cerebrovascular disease.

SECONDARY OUTCOMES:
Time to first coronary heart disease diagnosis | 52 weeks
  Analysed using Cox's proportional hazards model. Time from index smoking cessation attempt. Excluding patients with prior coronary heart disease.
Time to first cerebrovascular disease diagnosis | 52 weeks
  Analysed using Cox's proportional hazards model. Time from index smoking cessation attempt. Excluding patients with prior cerebrovascular disease.
Odds of recording one or more consultations for coronary heart disease or cerebrovascular disease | 52 weeks
  Analysed using conditional logistic regression model. Recorded General Practice consultations or hospital attendances for coronary heart disease or cerebrovascular disease, including General Practice consultations, Accident & Emergency attendance, out-patient department attendance or in-patient admissions.
Survival time for coronary heart disease-related death. | 52 weeks
  Analysed using Cox's proportional hazards model. Time from index smoking cessation attempt.
Survival time for cerebrovascular disease-related death. | 52 weeks
  Analysed using Cox's proportional hazards model. Time from index smoking cessation attempt.
Survival time for all-cause mortality. | 52 weeks
  Analysed using Cox's proportional hazards model. Time from index smoking cessation attempt.

OTHER OUTCOMES:
Survival time for coronary heart disease-related death | Any time after index smoking cessation attempt
  Analysed using Cox's proportional hazards model.
Survival time for cerebrovascular disease-related death | Any time after index smoking cessation attempt
  Analysed using Cox's proportional hazards model.
Survival time for all-cause mortality | Any time after index smoking cessation attempt
  Analysed using Cox's proportional hazards model.

CONTACTS AND LOCATIONS:
Overall Officials: David Price, Prof, MD, Principal Investigator — University of Aberdeen
Locations (1):
- Research in Real Life Ltd, Cambridge, United Kingdom

REFERENCES:
- [Background] Fiore MC, Bailey WC, Cohen SJ, et al. Treating tobacco use and dependence. Clinical practice guideline. Rockville (MD): US Department of Health and Human Services, Public Health Service, 2000
- [Background] West R, McNeill A, Raw M. Smoking cessation guidelines for health professionals: an update. Health Education Authority. Thorax. 2000 Dec;55(12):987-99. doi: 10.1136/thorax.55.12.987. PMID 11083883
- [Background] Le Foll B, George TP. Treatment of tobacco dependence: integrating recent progress into practice. CMAJ. 2007 Nov 20;177(11):1373-80. doi: 10.1503/cmaj.070627. PMID 18025429
- [Background] Stead LF, Perera R, Bullen C, Mant D, Lancaster T. Nicotine replacement therapy for smoking cessation. Cochrane Database Syst Rev. 2008 Jan 23;(1):CD000146. doi: 10.1002/14651858.CD000146.pub3. PMID 18253970
- [Background] Cahill K, Stead LF, Lancaster T. Nicotine receptor partial agonists for smoking cessation. Cochrane Database Syst Rev. 2007 Jan 24;(1):CD006103. doi: 10.1002/14651858.CD006103.pub2. PMID 17253581
- [Background] British Medical Association and the Royal Pharmaceutical Society of Great Britain. British National Formulary. Version 56. London; BNF Group; 2008.
- See also: World Health Organization (WHO). 2007. The European tobacco control report 2007 [online] — http://www.euro.who.int/__data/assets/pdf_file/0005/68117/E89842.pdf
- See also: eto R, Lopez AD, Boreham J, et al. 2006. Mortality from smoking in developed countries 1950 - 2000 (2nd ed.) [online] — http://www.deathsfromsmoking.net